CLINICAL TRIAL: NCT07254910
Title: Feasibility of a Multi-Channel Intervention to Promote Colorectal Cancer Screening Among American Indians in Oklahoma
Acronym: YVONNE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 16811
Record Dates: First submitted 2025-10-28; First posted 2025-11-28 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: CRC Screening; CRC (Colorectal Cancer)
Keywords: colorectal screening; virtual clinician; multi-channel communication; tribal outreach; Tribal Nations
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase 1: We will conduct 4 focus groups (n=6-8 per group) or individual interviews of AI patients from IHS Clinton Service Unit at the clinic or via Zoom. Groups will be stratified by past completion of previous FIT screening (yes/no) to compare perceived and structural barriers/facilitators to CRC screening. Intervention will be co-developed and employ value-centered design principles to tailor content to Cheyenne and Arapaho cultural norms. The CAB will be used to co-develop the focus group guides before use implementation with patients. Phase 2: The Tribal community health educator will be professionally recorded by the OU Health Marketing team to create Narrative Testimonial Video and v-TCHE interventions. The v-TCHE video will then be digitized to create a photorealistic v-TCHE will be created using the AI video generation system, Synethesia. Phase 3: Create a HIPAA-compliant, secure REDCap study database.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Narrative Testimonial Video of a Tribal Community Health Educator (Active Comparator): The narrative testimonial will provide a first-person recording of a real Tribal community health educator. In addition to the kernel information, the narrative video will employ culturally concordant storytelling about their personal experiences helping AI patients get screened and positive outcomes associated with early detection.
  Interventions: Behavioral: Narrative Testimonial Video
- v-TCHE Interaction (Active Comparator): Participants can interact via a set of authored responses or speak freely to the vTCHE. The v-TCHE uses Google Speech-to-Text to convert participant speech into text and Google's DialogFlow logs participants' selections, utterances, and interactions with the vTCHE. The interaction will elicit individual preferences, address concerns about CRC, and empower decision-making while still promoting CRC screening.
  Interventions: Behavioral: v-TCHE Interaction

INTERVENTIONS:
Behavioral: Narrative Testimonial Video — The narrative testimonial will provide a first-person recording of a real Tribal community health educator. In addition to the kernel information, the narrative video will employ culturally concordant storytelling about their personal experiences helping AI patients get screened and positive outcomes associated with early detection.
  Arms: Narrative Testimonial Video of a Tribal Community Health Educator
Behavioral: v-TCHE Interaction — Participants can interact via a set of authored responses or speak freely to the vTCHE. The v-TCHE uses Google Speech-to-Text to convert participant speech into text and Google's DialogFlow logs participants' selections, utterances, and interactions with the vTCHE. The interaction will elicit individual preferences, address concerns about CRC, and empower decision-making while still promoting CRC screening.
  Arms: v-TCHE Interaction

SUMMARY:
The Accelerating Colorectal Cancer Screening and follow-up through Implementation Science (ACCSIS) Program addresses major regional CRC screening disparities among AI in Oklahoma. The investigators are engaged in a participatory and collaborative effort with Tribal Nations, Area Indian Health Boards, and Indian Health Service (IHS) healthcare facilities. The overall objective of this proposal is to leverage these relationships and examine the feasibility of co-developing and disseminating a v-TCHE as part of a multi-channel communication intervention. To achieve this objective, the investigators have partnered with IHS Clinton Service Unit, which serves members of the Cheyenne and Arapaho Tribes. The intervention will be disseminated across two channels: (1) Social Media (i.e., accessed via online study adverts) and (2) Clinic (i.e., direct messaging to patients via a study link in a SMS text). Across both channels, the investigators will examine reach of the intervention and its potential efficacy via a randomized controlled trial. Once participants click on the study link they will be randomized 1:1 to one of two intervention conditions: (1) watch a Narrative Testimonial Video of a real-life Tribal community health educator (control) or (2) an interaction with a v-TCHE. Participants will then complete a post-intervention survey, in which they can click to order a FIT kit afterwards.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the second-leading cause of cancer death in both men and women in the United States.1 Compared to national averages, American Indians (AI) endure a disproportionate burden of CRC incidence and CRC-specific mortality.2 Screening is an effective early detection strategy to decrease preventable CRC-related deaths, but AI have some of the lowest CRC screening rates. In Oklahoma, only 51% of AI are up to date with screening compared to nearly two-thirds of eligible US adults.2 Efforts to improve screening rates have focused on increasing access to home stool screening (i.e.. fecal immunochemical test; FIT), as many AI live in rural communities and must drive long distances to access screening services. Tribal community health educators (TCHE) are an effective strategy to promote FIT screening within AI communities as they can overcome historical mistrust, health literacy gaps, and provide culturally concordant educational messaging. However, success of TCHE is limited by their reach as they cannot logistically engage with all necessary AI communities. As such, there remains a critical need to develop novel and scalable multi-channel communication interventions that can mimic the benefits of a TCHE and provide easy access to FIT kits among AI in Oklahoma. Virtual human technology, which uses 3D models to create photorealistic virtual humans, offers an innovative approach to create a virtual TCHE (v-TCHE) and may overcome the logistical barriers inherent with in-person delivered health education. The investigative team have previously used this technology to create race- and culturally concordant virtual characters to deliver CRC screening recommendations (R01CA207689) and support clinical trials enrollment (R24AG074867; U01CA274970) among rural and racial minority patients in Florida. This proposal would support codevelopment and testing of the first virtual human tailored for AI patients. The investigators believe a v-TCHE can engender the positive source cues that invoke feelings of trust among AI patients that an in-person TCHE provides. The novelty and customization of a v-TCHE can further enhance interest and perceived cultural relevance of CRC screening information. Moreover, the interactive nature, compared to other more passive communication strategies (e.g., narrative testimonial videos), can empower decisionIRB NUMBER: 16811 IRB APPROVAL DATE: 04/10/2024 Neil, Version # IRB version 03/12/2019 3 making and aligns with cultural preference of self-determination within Tribal practices while still promoting CRC screening.3 Aim 1. Co-develop a multi-channel communication intervention with AI in Oklahoma. Approach. Phase 1 will conduct 4 focus groups (n=6-8 per group) of AI patients from IHS Clinton Service Unit to co-develop the communication intervention content. Phase 2 will record the Narrative Testimonial Video and create the v-TCHE. Phase 3 will employ a community advisory board (CAB) for final review of the interventions before dissemination. Aim 2. Determine the reach and potential efficacy of a multi-channel communication intervention to promote CRC screening among AI in Oklahoma. Approach. The investigators aim to accrue 150 AI patients, aged 45-75 and not up to date with CRC screening, who live within IHS Clinton Service Unit catchment area. Reach (primary outcome) will be determined by the proportion of participants who successfully engage with the intervention, compared across intervention channels (Social Media vs. Clinic). Potential efficacy will be determined by (1) post-intervention differences in knowledge about CRC symptoms and screening and (2) the proportion of participants who order and return a FIT kit within 30 days, compared between study conditions (i.e., Narrative Testimonial Video vs. v-TCHE interaction) and intervention channels (Social Media vs. Clinic). Public Health Impact. This proposal is highly responsive to Track 2 in the PA-20-272 as it attempts to address inequities in CRC outcomes among AI populations. The investigators examine the feasibility of co-developing and disseminating a multi-channel communication intervention to promote a United States Preventive Services Taskforce recommended cancer screening test. If successful, findings will support a first-of-its-kind, highly scalable approach to overcome the reach limitations that Tribal community health educators face. A future R01 will determine the efficacy of different v-TCHE to promote FIT screening across other Tribal healthcare systems.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-75 Live within IHS Clinton Service Unit catchment area Fluent in English and read at or above 6th grade level Self report as American Indian or have CDIB

Exclusion Criteria:

* Self report up to date with CRC screening FIT within 1 year

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Reach | From enrollment to the end of the intervention at 30 days
  The percentage of participants who successfully engage with the intervention (i.e., via click through rate) and compared across intervention channels (Social Media vs. Clinic). A GIS analysis will determine where reach was geographically greatest.

SECONDARY OUTCOMES:
Potential efficacy | From enrollment to the end of intervention at 30 days
  Participants will complete minimal survey assessments for study intervention. Post-intervention survey measures will be limited to multi-dimensional objective assessments of knowledge about CRC and screening, confidence in identifying CRC symptoms, key theoretical constructs associated with CRC screening (e.g., self-efficacy, response efficacy), and intervention evaluation (e.g., acceptability, cultural appropriateness).
FIT Kit Screening | 30 days
  The proportion of participants who order and return a FIT kit within 30 days, compared between intervention conditions (i.e., Narrative Testimonial Video vs. v-TCHE interaction) and intervention channels (Social Media vs. Clinic). Participants who return a FIT kit and report an abnormal finding, will be provided multiple forms of navigation to support follow-up care, including SMS text message/email and phone calls from study and clinic navigators.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Neil, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- TSET Health Promotion Research Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
Research analysis will only be conducted by IRB-approved key study personnel. No de-identified individual participant data will be shared outside the primary research group.